CLINICAL TRIAL: NCT03905746
Title: Expression and Variance of microRNAs in a Cohort of Patients With Acute Decompensation of Cirrhosis.
Brief Title: Study of microRNAs in a Decompensated Cirrhosis
Acronym: EmiC
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0020; 2019-A00266-51 (Other: ID-RCB)
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Cirrhosis; Acute Decompensation
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and peripheral blood mononuclear cells (PBMCs) will be collected at D0, D2 and D7 from enrolment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- acute decompensation group: patients admitted within 48 hours for acute decompensation of cirrhosis, with or without evidence of sepsis
  Interventions: Other: blood sample at Day 0; Other: blood sample at Day 2 and Day 7; Other: stool sample at Day 0
- Pathological control group: patients with Chronic Liver Disease (CLD), also named stable cirrhotic patients, without any admission in the last 6 months for an acute event
  Interventions: Other: blood sample at Day 0; Other: stool sample at Day 0

INTERVENTIONS:
Other: blood sample at Day 0 — 40mL blood (plasma and PBMCs) will be performed at D0 (inclusion), at the time of routine exams.
  (20 ml will be used for study analyzes ; 20mL will constitute the biological collection)
Other: blood sample at Day 2 and Day 7 — 20mL blood (plasma and PBMCs) will be performed at Day 2 and Day 7 from recruitment, at the time of routine exams. These two samples will constitute the biological collection.
  Groups: acute decompensation group
Other: stool sample at Day 0 — stool sample (2mL) will be performed at D0 (inclusion), at the time of routine exams.

SUMMARY:
Cirrhotic patients are at higher risk of sepsis due to impaired innate and adaptive immune responses. Septic complications represent a major issue in the management of cirrhotic patients, with a 1-month mortality rate of 23%, which increases to 80% at 3 months in case of associated organ failure.

Delay to treatment initiation during a septic episode may increase the risk of complications and mortality of cirrhotic patients. However, the inappropriate use of antibiotics exposes cirrhotic patients to the risk of more severe infections due to multi-resistant organisms or fungi.

The use of diagnostic markers for sepsis is limited in the context of cirrhosis because of the lack of hepatic synthesis of these markers on the one hand and non-specific inflammation related to cirrhosis on the other hand.

Therefore, it is necessary to develop new tools for the early diagnosis of sepsis and appropriate management of cirrhotic patients.

The interest of microRNAs (miRNAs) in the diagnosis and prognosis of septic shock has been reported in the general population. No studies have described circulating miRNAs or reported their interest in the diagnosis of sepsis in a population of cirrhotic patients with acute decompensation (AD).

This preliminary study of 800 circulating miRNAs will be performed in a cohort of patients with acute cirrhosis decompensation, for whom the incidence of sepsis is estimated at 40%. The aim to evaluate the interest and feasibility of a larger study on the interest of circulating miRNAs in the early diagnosis of sepsis in cirrhotic patients. The long-term objective of this study is the development of biomarkers for the early management of cirrhotic patients with sepsis and the rationalization of antibiotic use to improve their prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis (determined either by histopathology or by association of clinical signs of portal hypertension and hepatocellular insufficiency and radiological signs (dysmorphic liver, evidences of portal hypertension (collateral circulation, ascites)).

AND

* Not refusing his / her participation in the study after information (or non-opposition of the person of confidence if the patient has a disorder of consciousness or impaired judgment (hepatic encephalopathy) at the time of inclusion) AND
* Admitted within 48 hours for an episode of acute decompensation (acute decompensation group = AD group), which is defined by the sudden occurrence of one or more of the following clinical or biological symptoms:

  * Jaundice
  * Hepatic encephalopathy
  * oedemato-ascitic decompensation
  * Gastro-intestinal bleeding
  * Acute renal failure (according to AKIN criteria (22)) and / or hyponatremia
  * Degradation of hepatocellular functions (decrease of prothrombin time and factor V measured in blood, increase of bilirubinemia) OR
* Outpatient follow-up for stable cirrhosis, not admitted in the last 6 months for an episode of acute cirrhosis decompensation (pathological control group)

Exclusion Criteria:

* Minor or major patient under guardianship or curatorship
* Pregnant women
* Patient deprived of liberty
* History of extra-digestive cancer
* History of hepatocellular carcinoma or other hepatobiliary cancer
* Chronic infection with Hepatitis B virus (defined by the presence of Antibodies to hepatitis B core antigen (anti-HBc) and the absence of Hepatitis B surface antibodies (anti-HBs)) identified by a recent serology (less than 6 months)
* Chronic Hepatitis C Virus infection or cured for less than 6 months
* Infection with the Human Immunodeficiency Virus identified by a recent serology (less than 6 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients concerned are cirrhotic patients, followed in the hepatology department of Pr Zoulim, in gastroenterology department of Dr Marielle Guillet and in intensive care unit of Dr Céline Guichon (Croix Rousse Hospital, North Hospital Group, Hospices Civils de Lyon), without a history of cancer or active infection with the virus of the hepatitis B, hepatitis C virus or HIV.
  2 groups will be formed:
  * A group of cirrhotic patients with acute decompensation (AD group)
  * A group of stable cirrhotic patients (pathological controls)
Sampling Method: Non-Probability Sample
Enrollment: 444 (Estimated)
Dates: Start 2019-06-26 (Actual); Primary Completion 2033-12-26 (Estimated); Study Completion 2034-06-26 (Estimated)

PRIMARY OUTCOMES:
Plasma levels of 800 miRNA between the 2 subgroups of the AD group according to the retrospective diagnosis of sepsis or not | Day 0
  The difference of miRNAs levels will assess in patients recruited in the AD group who will be retrospectively diagnosed as septic at the time of enrollment and compare them non septic patients.

SECONDARY OUTCOMES:
miRNA profiles | Day 0
  Difference between miRNA profiles identified in a subgroup of patients with secondary infection during admission (DA group) and a subgroup of patients who did not developing a secondary infection on admission
miRNA profiles | Day 2
  Difference between miRNA profiles identified in a subgroup of patients with secondary infection during admission (DA group) and a subgroup of patients who did not developing a secondary infection on admission
miRNA profiles | Day 7
  Difference between miRNA profiles identified in a subgroup of patients with secondary infection during admission (DA group) and a subgroup of patients who did not developing a secondary infection on admission
miRNA profiles | Day 0
  Difference in miRNA profiles identified in a subgroup of patients with secondary infection 6 months, 1 year and 6 years after inclusion (DA group) and a subgroup of patients developing no secondary infection during follow-up (DA group).
miRNA profiles | Day 2
  Difference in miRNA profiles identified in a subgroup of patients with secondary infection 6 months, 1 year and 6 years after inclusion (DA group) and a subgroup of patients developing no secondary infection during follow-up (DA group).
miRNA profiles | Day 7
  Difference in miRNA profiles identified in a subgroup of patients with secondary infection 6 months, 1 year and 6 years after inclusion (DA group) and a subgroup of patients developing no secondary infection during follow-up (DA group).
Correlation between plasma levels of 800 miRNAs and degree of portal hypertension | Day 0
Correlation between plasma levels of 800 miRNAs and nutritional profile (Liver Frailty Index, bracchial circumference) | Day 0
miRNA profiles | Day 0
  Difference between miRNA profiles identified in different subgroups of patients in the DA group according to the mode progression (PREDICT study criteria)
miRNA profiles | Day 2
  Difference between miRNA profiles identified in different subgroups of patients in the DA group according to the mode progression (PREDICT study criteria)
miRNA profiles | Day 7
  Difference between miRNA profiles identified in different subgroups of patients in the DA group according to the mode progression (PREDICT study criteria)
Correlation between monocyte expression of HLA-DR (mHLA-DR) and circulating miRNA expression | Day 0
Correlation between monocyte expression of HLA-DR (mHLA-DR) and circulating miRNA expression | Day 2
Difference in miRNA profiles between patients who died without liver transplantation at 6 months, 1 year and 5 years from inclusion and surviving patients. | Day 0
  DA group and pathological control
Difference in miRNA profiles between patients who died without liver transplantation at 6 months, 1 year and 5 years from inclusion and surviving patients. | Day 2
  DA group
Difference in miRNA profiles between patients who died without liver transplantation at 6 months, 1 year and 5 years from inclusion and surviving patients. | Day 7
  DA group
Difference in miRNA profiles between patients with a new episode of cirrhosis decompensation at 6 months, 1 year and 5 years from inclusion and surviving patients (DA group) | Day 0
  DA group
Difference in miRNA profiles between patients with a new episode of cirrhosis decompensation at 6 months, 1 year and 5 years from inclusion and surviving patients (DA group) | Day 2
  DA group
Difference in miRNA profiles between patients with a new episode of cirrhosis decompensation at 6 months, 1 year and 5 years from inclusion and surviving patients (DA group) | Day 7
  DA group
Difference between miRNA profiles / subgroup of the pathological control group presenting a 1st episode of cirrhosis decompensation and in the subgroup presenting no 1st episode of cirrhosis decompensation at 6 months, 1 and 5 years of inclusion | Day 0
  pathological control group
Association between miRNA expression and PBMC phenotype in the different groups (DA and pathological controls) and subgroups | Day 0
  control group and DA group / Subgroups :DA group: infection or not, secondary infection or not, evolutionary profile; pathological control group: decompensation at 6 Months, 1 and 5 years or not
Association between miRNA expression and PBMC phenotype in subgroups (DA group: infection or not, secondary infection or not, evolutionary profile at 6 Months, 1 year and 5 years or not) | Day 2
  DA group
Association between miRNA expression and PBMC phenotype in subgroups (DA group: infection or not, secondary infection or not, evolutionary profile at 6 Months, 1 year and 5 years or not) | Day 7
  DA group
Phenotypic and functional profiles of T and B lymphocytes from patients with cirrhosis at different stages (pathological control group and DA group) | Day 0
  pathological control group and DA group ; determined by spectral cytometry on the one hand, and single cell RNA sequencing and single cell secretome analysis on the other.
Phenotypic and functional profiles of T and B lymphocytes from patients with cirrhosis at different stages (pathological control group and DA group) | Day 2
  DA group ; determined by spectral cytometry on the one hand, and single cell RNA sequencing and single cell secretome analysis on the other.
Phenotypic and functional profiles of T and B lymphocytes from patients with cirrhosis at different stages (pathological control group and DA group) | Day 7
  DA group ; determined by spectral cytometry on the one hand, and single cell RNA sequencing and single cell secretome analysis on the other.
Predictive value of miRNAs, ADM and cDPP3 for risk of secondary infection, further decompensation, death without liver transplantation. | Day 0
  control group and DA group ; Predictive value will be assessed by ROC curve ant AUC and then logistic regression will be performed.
Predictive value of miRNAs, ADM and cDPP3 for risk of secondary infection, further decompensation, death without liver transplantation. | Day 2
  DA group ; Predictive value will be assessed by ROC curve ant AUC and then logistic regression will be performed.
Predictive value of miRNAs, ADM and cDPP3 for risk of secondary infection, further decompensation, death without liver transplantation. | Day 7
  DA group ; Predictive value will be assessed by ROC curve ant AUC and then logistic regression will be performed.
Correlation between i) the proportion of T and B cells circulating subpopulations and ii) circulating levels of potential biomarkers (concentrations of cytokines in plasma, concentration of circulating bacterial DNA). | Day 0
  control group and DA group
Correlation between i) the proportion of T and B cells circulating subpopulations and ii) circulating levels of potential biomarkers (concentrations of cytokines in plasma, concentration of circulating bacterial DNA). | Day 2
  DA group
Correlation between i) the proportion of T and B cells circulating subpopulations and ii) circulating levels of potential biomarkers (concentrations of cytokines in plasma, concentration of circulating bacterial DNA). | Day 7
  DA group

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de la Croix Rousse, Lyon, France